CLINICAL TRIAL: NCT05514574
Title: The Effect of Listening to Music and Stress Ball Application on Patients' Anxiety Level and Hemodynamic Parameters During Percutaneous Coronary Intervention
Brief Title: The Effect of Listening to Music and Stress Ball Application on Patients' Anxiety Level and Hemodynamic Parameters During PCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keriman Yildiz (Other)
Collaborators: Necmettin Erbakan University (Other)
Responsible Party: Sponsor-Investigator, Keriman Yildiz, Study Director, Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KYildiz
Record Dates: First submitted 2022-08-17; First posted 2022-08-24 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Percutaneous Coronary Intervention; Anxiety; Hemodynamics
Keywords: percutaneous coronary intervention; anxiety; hemodynamics; music; stress ball
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Prospective Non-Randomized Controlled Clinical Trial
Who Masked: Outcomes Assessor
Masking Description: Patients and their relatives, clinical staff, will be blinded to the group assignment. Evaluation of the data will be done by a blinded technique by a biostatistician not involved in the study and blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music (Experimental): Patients (listening to music group) who are taken to the intervention table and placed on their backs by the team that will perform the intervention will be monitored. The hemodynamic parameters on the monitor screen will be recorded on the data collection form before and after percutaneous coronary intervention by the researcher KY. Anxiety levels of patients will be evaluated by the researcher KY with the State Anxiety Scale before being taken to the intervention room for percutaneous coronary intervention (while in a bed or stretcher or wheelchair). Anxiety levels of patients will be evaluated by the researcher KY with the State Anxiety Scale after leaving the intervention room (while on the bed or stretcher). During percutaneous coronary intervention; Except for routine treatment and care interventions, the patient will listen to music during the procedure.
  Interventions: Other: Music
- Stress ball (Experimental): Patients (stress ball group) who are taken to the intervention table and placed on their backs by the team that will perform the intervention will be monitored. The hemodynamic parameters on the monitor screen will be recorded on the data collection form before and after percutaneous coronary intervention by the researcher KY. Anxiety levels of patients will be evaluated by the researcher KY with the State Anxiety Scale before being taken to the intervention room for percutaneous coronary intervention (while in a bed or stretcher or wheelchair). Anxiety levels of patients will be evaluated by the researcher KY with the State Anxiety Scale after leaving the intervention room (while on the bed or stretcher). During percutaneous coronary intervention; Except for routine treatment and care interventions, the patient will stress ball will be applied during the procedure.
  Interventions: Other: Stress ball
- Control (No Intervention): Patients (control group) who are taken to the intervention table and placed on their backs by the team that will perform the intervention will be monitored. The hemodynamic parameters on the monitor screen will be recorded on the data collection form before and after percutaneous coronary intervention by the researcher KY. Anxiety levels of patients will be evaluated by the researcher KY with the State Anxiety Scale before being taken to the intervention room for percutaneous coronary intervention (while in a bed or stretcher or wheelchair). Anxiety levels of patients will be evaluated by the researcher KY with the State Anxiety Scale after leaving the intervention room (while on the bed or stretcher). During percutaneous coronary intervention; No intervention will be performed except for routine treatment and care interventions.

INTERVENTIONS:
Other: Music — "hussoni duseni " music
  Arms: Music
Other: Stress ball — Stress ball squeeze
  Arms: Stress ball

SUMMARY:
In this study, it was aimed to determine the effects of listening to music and applying a stress ball on patients' anxiety level and hemodynamic parameters during percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Percutaneous coronary intervention causes patients to experience anxiety and change their hemodynamic parameters. In this study, it was aimed to determine the effects of listening to music and applying a stress ball on patients' anxiety level and hemodynamic parameters during percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older,
* Literate,
* Able to communicate verbally,
* Turkish speaking,
* No hearing or vision loss,
* No sensory or motor deficits in the hand or arm,
* Percutaneous coronary intervention will be applied,
* intervention from the femoral artery,
* Voluntarily participated in the research,
* Patients signing the informed consent form will be included.

Exclusion Criteria:

* Under the age of 18,
* Not signing the informed consent form,
* Illiterate,
* Unable to speak Turkish,
* Unable to communicate verbally
* Those who have a neurological or psychiatric disease that prevents communication,
* Hearing and sight impaired,
* Those who have had a mastectomy
* Those with arterio-venous fistula
* Percutaneous coronary intervention has been performed in the last 2 years,
* Restricted special groups (pregnant women, criminal convicts, etc.),
* Emergency cases where communication cannot be established,
* Those with equipment problems such as monitors and cuffs,
* Those who will be given sedatives during the procedure,
* Those who will be taking cardiovascular system medications other than routine practices during the procedure,
* Those who will be given oxygen during the procedure,
* Patients who are treated from a different artery other than the femoral artery will not be accepted.

Criteria for exclusion from follow-up:

* Those who want to quit working,
* Those who give up listening to music,
* Those who give up using the stress ball,
* Those who were given cardiovascular system medications other than routine practices during the procedure,
* Those who underwent intervention from a different artery instead of the femoral artery,
* Those who do not want to wear headphones because they cannot hear the doctor's questions
* Those whose second measurements could not be taken because they were quickly removed from the interventional room,
* Those who underwent carotid artery angiography in addition to coronary artery,
* Those who give incorrect PCI history,
* Those who cannot listen to music or whose music is interrupted due to connection problems,
* Those whose intervention cannot be performed at the planned time due to urgent patient arrival,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
State Anxiety Score | Each participant's State Anxiety score will be measured before and after admission to (twice-daily) the percutaneous coronary intervention room will be followed for 1 day (day of the attempt) will be recorded in the data collection form.
  Change in State Anxiety Score after intervention.

SECONDARY OUTCOMES:
Systolic Blood Pressure Value (mmHg) | Systolic Blood Pressure value of each participant will be measured in the pre- and post-procedure (twice-daily) in percutaneous coronary intervention room will be followed for 1 day (day of the attempt) will be recorded in the data collection form
  Change in Systolic Blood Pressure Value after intervention.
Diastolic Blood Pressure Value (mmHg) | Diastolic Blood Pressure value of each participant will be measured in the pre- and post-procedure (twice-daily) in percutaneous coronary intervention room will be followed for 1 day (day of the attempt) will be recorded in the data collection form.
  Change in Diastolic Blood Pressure Value after intervention.
Mean Arterial Pressure Value (mmHg) | Mean Arterial Pressure value of each participant will be measured in the pre- and post-procedure (twice-daily) in percutaneous coronary intervention room will be followed for 1 day (day of the attempt) will be recorded in the data collection form.
  Change in Mean Arterial Pressure Value after intervention.
Heart Rate/Minute Value | Heart Rate/Minute value of each participant will be measured in the pre- and post-procedure (twice-daily) in percutaneous coronary intervention room will be followed for 1 day (day of the attempt) will be recorded in the data collection form.
  Change in Heart Rate/Minute Value after intervention.
Respiratory Rate/Minute Value | Respiratory Rate/Minute value of each participant will be measured in the pre- and post-procedure (twice-daily) in percutaneous coronary intervention room will be followed for 1 day (day of the attempt) will be recorded in the data collection form.
  Change in Respiratory Rate/Minute Value after intervention.
Peripheral Oxygen Saturation (SpO2) Value | Peripheral Oxygen Saturation value of each participant will be measured in the pre- and post-procedure (twice-daily) in percutaneous coronary intervention room will be followed for 1 day (day of the attempt) will be recorded in the data collection form.
  Change in Peripheral Oxygen Saturation Value after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: SERPİL YÜKSEL, PhD, Principal Investigator — Necmettin Erbakan University; AHMET YILMAZ, PhD, Study Director — Karamanoğlu Mehmetbey University; KERİMAN YILDIZ, MSc, Study Director — Necmettin Erbakan University
Locations (1):
- Karaman Provincial Health Directorate Karamanoğlu Mehmetbey University Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
STUDY PROTOCOL
Supporting Information: Study Protocol
Time Frame: After December 1, 2024
Access Criteria: Anyone who wishes to access the data. Study Protocol.